CLINICAL TRIAL: NCT06167590
Title: Integrins and Protocadherins in Glutamatergic Circuits: Identification of Common Signaling Pathways and Molecular Targets in Anxiety and Major Depressive Disorders (GAPsy)
Acronym: GAPsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: CNR Institute of Neuroscience, Parma (Other); University of Trieste (Other); IRCCS Fondazione Stella Maris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GAPsy
Record Dates: First submitted 2023-05-22; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-05

CONDITIONS: Depression, Anxiety; Healthy
Keywords: Depression, Anxiety; Healthy controls; Neuroimaging; Functional magnetic resonance imaging (fMRI); Proton magnetic resonance spectroscopy (1H-MRS); Murine models; Integrin β3; Protocadherin 9; CRISPR-mediated transcription activation (CRISPRa)
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anxious-depressive disorder (Other)
  Interventions: Diagnostic Test: GAPsy protocol
- Healthy controls (Other)
  Interventions: Diagnostic Test: GAPsy protocol

INTERVENTIONS:
Diagnostic Test: GAPsy protocol — Each participant will undergo a 7 T multimodal neuroimaging session, including T1-weighted, 1H-MRS and fMRI. Each participant will also be assessed through a structured clinical interview (SCID-I e SCID-II) and will be administered scales such as HAM-A, HAM-D, BPRS and MADRS.

SUMMARY:
The aim of this study is to identify biologically viable targets for the treatment of major depressive disorder (MDD) and anxiety disorder (AD) with the ultimate goal of guiding physicians' therapeutic strategies and identifying more effective and safer treatments for patients. Following the inclusion and exclusion criteria, the investigators will recruit 10 patients with a diagnosis of anxious-depressive disorder (MDD-AD) and 10 healthy controls (HC) subjects. Each participant will be evaluated by a team of expert psychologists and physicians, who will be conducting a structured interview and administering a set of psychopathological scales to assess the symptoms' severity. The participants will also undergo7T multimodal neuroimaging session (including T1-weighted, 1H-MRS and fMRI).

In the second part of the study, murine models will be used to study the role of integrin β3 (Itgb3) and protocadherin 9 (Pcdh9) in glutamatergic transmission at a molecular level and to evaluate whether the electrophysiological and behavioral defects identified in Itgb3- and Pcdh9-knockout mice can be restored by CRISPR-mediated transcription activation (CRISPRa).

DETAILED DESCRIPTION:
The study is structured into two parts. In the first part the investigators will be recruiting 10 patients with MDD-AD and 10 HC, following the inclusion and exclusion criteria. Each participant will be evaluated by a team of experienced psychologists and clinicians, administering structured clinical interviews to assess the presence/absence of axis I and II psychiatric disorders (SCID-I and SCID-II) (first visit). Furthermore, in all subjects the degree of depressive/manic dysintomatology will be measured through the use of clinical scales and psychopathological tests such as:the Hamilton Depression Rating Scale (HAM-D), the Montgomery- Asberg Depression rating Scale (MADRS), the Hamilton Anxiety Rating Scale (HAM-A) and the Brief Psychiatric Rating Scale (BPRS)(second visit; within one week of the first screening visit). Moreover, additional clinical data will beextrapolated from medical records and interviews with psychiatrists (if available).

The investigators will also evaluate the suitability of each participant to undergo the multimodal acquisition of Magnetic Resonance Imaging (MRI) data with a 7T GE scanner. The neuroimaging session, performed during the third visit (within one month of the second visit) will include:

* T1-weighted image acquisition: to study the volumetric differences of white and gray matter between subjects in the prefrontal-limbic pathway.
* fMRI: to assess functional connections between prefrontal cortex and limbic system.
* 1H-MRS: to study glutamatergic neurotransmission within the anterior cingulate and dorsolateral prefrontal cortex.

The sequences will be optimized thanks to the 32-channel brain coil (NovaMedical), to reduce artifacts and inhomogeneities in images.

The second part of the study will involve murine models. More specifically, to assess whether Pcdh9 deficits affect the number and morphology of excitatory synapses, electron microscopic analyses will be performed in Pcdh9-knockout mice. Glutamatergic signaling will also be studied at the biochemical level: the expression levels of all major glutamate receptor subunits (ionotropic and metabotropic) will be investigated by analyzing cortical protein lysates (total lysates) in adult mice (3-4 months). In addition, to identify finer changes in glutamate receptor expression, their intracellular and surface expression will be analyzed using the BS3 crosslinking assay.

The investigators will also proceed in the characterization of the interaction between integrin β3 and Protocadherin9 using co-immunoprecipitation analysis from mouse brain: in case of positive results (at least 3 replicates), further analysis will be conducted to study whether the two proteins bind directly.

Electrophysiological characterization of Itgb3 and Pcdh9 murine patterns in the medial prefrontal cortex at both synaptic and local network levels will also be performed and, lastly, an evaluation of functional recovery of behavioral and electrophysiological deficits mediated by CRISPRa will be conducted. In this case, experiments on murine models will be perform to determine whether overexpression of integrin β3 or protocadherin9 could compensate for defects in synaptic glutamatergic transmission caused by deficiencies in CAMs.

ELIGIBILITY:
Inclusion Criteria:

* Patients group: diagnosis of anxiety-depressive disorder based on the DSM-5 diagnostic criteria; age range between 18 and 35 years; age of onset < 2 years; severe or moderate depression based on scores on the Hamilton Depressive Rating Scale (HAM-D; scores between 14 and 24); severe or moderate anxiety based on scores on the Hamilton Anxiety Rating Scale (HAM-A; scores between 18 and 30); patients must have both severe/moderate depression and anxiety to be included; ability and willingness to provide informed consent and adhere to study procedures.
* Healthy controls group: age range between 18 and 35 years; ability and willingness to provide informed consent and adhere to study procedures.

Exclusion Criteria:

* Patients group: diagnosis of other Axis I and/or Axis II psychiatric conditions; substance and/or alcohol abuse and/or dependence; tumors or liver disorders; cognitive impairment.
* Healthy controls: history of Axis I psychiatric conditions in first-degree relatives; presence of preexisting neurological conditions; substance and/or alcohol abuse and/or dependence; cognitive impairment.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-07-14 (Estimated); Study Completion 2025-07-14 (Estimated)

PRIMARY OUTCOMES:
Brain structure differences in terms of white matter in the prefrontal-limbic pathway | At T2 (third visit, within a month from the second visit)
  Evaluation of volumetric differences in terms of white matter in the prefrontal-limbic pathway, comparing the healthy controls group and the patients group, using structural neuroimaging (MRI)
Brain structure differences in terms of gray matter in the prefrontal-limbic pathway | At T2 (third visit, within a month from the second visit)
  Evaluation of volumetric differences in terms of white matter in the prefrontal-limbic pathway, comparing the healthy controls group and the patients group, using structural neuroimaging (MRI)
Functional connectivity differences in the prefrontal-limbic pathway | At T2 (third visit, within a month from the second visit)
  Evaluation of connectivity differences at rest and during task in the prefrontal-limbic pathway, comparing the healthy controls group and the patients group, using functional neuroimaging (fMRI)
Differences in the glutamatergic neurotransmission in the anterior cingulate and prefrontal dorsolateral cortices as assessed by using 1H-MRS | At T2 (third visit, within a month from the second visit)
  Evaluation of glutamatergic neurotransmission differences in the anterior cingulate and prefrontal dorsolateral cortices, comparing the healthy controls group and the patients group, using in vivo proton magnetic resonance spectroscopy (1H-MRS)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Maria Pozzoli, PhD, Principal Investigator — S. C. Psichiatria - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, MI, Italy

REFERENCES:
- [Background] Gorwood P. Generalized anxiety disorder and major depressive disorder comorbidity: an example of genetic pleiotropy? Eur Psychiatry. 2004 Feb;19(1):27-33. doi: 10.1016/j.eurpsy.2003.10.002. PMID 14969778
- [Background] Zhou Y, Cao Z, Yang M, Xi X, Guo Y, Fang M, Cheng L, Du Y. Comorbid generalized anxiety disorder and its association with quality of life in patients with major depressive disorder. Sci Rep. 2017 Jan 18;7:40511. doi: 10.1038/srep40511. PMID 28098176
- [Background] Jaso BA, Niciu MJ, Iadarola ND, Lally N, Richards EM, Park M, Ballard ED, Nugent AC, Machado-Vieira R, Zarate CA. Therapeutic Modulation of Glutamate Receptors in Major Depressive Disorder. Curr Neuropharmacol. 2017;15(1):57-70. doi: 10.2174/1570159x14666160321123221. PMID 26997505
- [Background] Abdallah CG, Jiang L, De Feyter HM, Fasula M, Krystal JH, Rothman DL, Mason GF, Sanacora G. Glutamate metabolism in major depressive disorder. Am J Psychiatry. 2014 Dec 1;171(12):1320-7. doi: 10.1176/appi.ajp.2014.14010067. Epub 2014 Oct 31. PMID 25073688
- [Background] Hastings RS, Parsey RV, Oquendo MA, Arango V, Mann JJ. Volumetric analysis of the prefrontal cortex, amygdala, and hippocampus in major depression. Neuropsychopharmacology. 2004 May;29(5):952-9. doi: 10.1038/sj.npp.1300371. PMID 14997169